CLINICAL TRIAL: NCT01794962
Title: Classification Based "Cognitive Functional Therapy" vs. Manual Therapy for a Subgroup of Patients With Chronic NSLBP, Classified as Having a "Flexion Pattern"
Brief Title: "Cognitive Functional Therapy" vs. Manual Therapy for Non-specific Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KU2012
Record Dates: First submitted 2013-01-27; First posted 2013-02-20 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain
Keywords: Classification; LBP; Cognitive functional therapy; Manual Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual therapy and exercises (Experimental): Manual therapy treatment: spinal manipulation, Soft tissue treatment, muscle energy techniques. Exercises: stabilisation exercises, Mckenzie exercises and general muscle exercises.
  Interventions: Other: manual therapy and exercises
- Cognitive Functional Therapy (Experimental): An in depth interview, including investigating the patients beliefs on back pain, fear towards movement, anxiety and distress, using reflecting questions. The physical part consists of specific and functional exercises related to the patients functional complaints.And general physical activity for 30 mins 3-4 times weekly.
  Interventions: Other: Cognitive functional therapy

INTERVENTIONS:
Other: Cognitive functional therapy — The intervention is directed at the maladaptive cognitive, physical and lifestyle behaviours associated with the disorder.
  Arms: Cognitive Functional Therapy
Other: manual therapy and exercises — Patients in this group will be treated with joint mobilization or manipulation techniques applied to the spine or pelvis primarily and is designed to be consistent with best current manual therapy practice.
  Arms: Manual therapy and exercises

SUMMARY:
This is a pilot study. Chronic LBP is a major health care problem in Denmark. Few patients receive a specific diagnosis, leaving the majority of patients diagnosed with non specific low back pain(NSLBP). Classification systems can help to guide the treatment of NSLBP. This pilot study will compare manual therapy (manipulation and soft tissue treatment)and exercises to a classification based biopsychosocial intervention (a cognitive/functional approach) as described by Peter O'Sullivan, on a subgroup called "flexion pattern"

This pilot study has three specific aims:

(i) To determine the mean and standard deviation on the numerical rating scale of participants in this setting who have a motor control flexion pattern, so that sample size calculations for a fully powered randomized controlled trial could be performed.

(ii) To test the logistical and practical procedures that will be required to perform a fully powered randomized controlled trial using these two treatments.

(iii) To gain a preliminary estimate of any difference in the effect of these two treatments, so as to determine if the results of a fully powered randomized controlled trial might be clinically important and therefore worthwhile undertaking

DETAILED DESCRIPTION:
This is a pilot study. Chronic LBP is a major health care problem in Denmark. Few patients receive a specific diagnosis, leaving the majority of patients diagnosed with non specific low back pain(NSLBP). Classification systems can help to guide the treatment of NSLBP.This project will recruit patients , classified with a "flexion pattern" according to the classification system proposed by Peter O´Sullivan. When classified with a flexion pattern the patients will be randomized into either of two treatment arms. Manual therapy (manipulation and soft tissue treatment)and exercises by a chiropractor or to a classification based biopsychosocial intervention done by a physiotherapist, (a cognitive/functional approach) as described by Peter O'Sullivan

This pilot study has three specific aims:

(i) To determine the mean and standard deviation on the numerical rating scale of participants in this setting who have a motor control flexion pattern, so that sample size calculations for a fully powered randomized controlled trial could be performed.

(ii) To test the logistical and practical procedures that will be required to perform a fully powered randomized controlled trial using these two treatments.

(iii) To gain a preliminary estimate of any difference in the effect of these two treatments, so as to determine if the results of a fully powered randomized controlled trial might be clinically important and therefore worthwhile undertaking

ELIGIBILITY:
Inclusion Criteria:

Participants must be between 18 - 65 years old and have, with a history of low back pain more than three months.

The primary pain area from T12- to the gluteal folds. Low back pain must be provoked by movements and/or physical activities. Average pain intensity in the last two weeks must be al least: 4/10 on Pain numerical rating scale Participants must have adequate comprehension and expressing the Danish language.

Participants must be classified as having a "flexion pattern".

Exclusion Criteria:

Participants must not have been sick listed for more than 4 months; have an acute exacerbation of LBP, surgery of low limb within last 4 months or hip or knee osteoarthritis limiting loading of knee and hip flexion.

Follow medical conditions are also excluding participants:

A history of spinal surgery Radicular pain (disc prolapse or foraminal stenosis): non painful symptoms in leg, clinical signs of altered nerve conduction) Spinal stenosis A previous history psychiatric disease Current pregnancy Widespread non-specific pain (for filling criteria for fibromyalgia) Imaging confirming spondylolisthesis

Other diseases:

Rheumatoid arthritis ankylosing spondylitis neurologic disease infection cancer previous history of osteoporosis The patient can´t be classified as having a flexion pattern Lack of compliance during the intervention: if a patient fails to turn up for more than one appointment with out prior notice.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity(numerical rating scale) | 12 months FU
  Pain intensity Numerical Rating Scale, as pain is the primary reason for patients to seek care. Numerical Rating Scales have shown to have reliability, validity and responsiveness to change at a best practise standard.

SECONDARY OUTCOMES:
Ronald Morris Questionaire | 12 months follow up

OTHER OUTCOMES:
Fear/Avoidance Beliefs Questionaire | 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Ussing, Msc, Principal Investigator — Spine Centre of Southern Denmark
Locations (1):
- Kasper Ussing, Middelfart, Fyn, Denmark